CLINICAL TRIAL: NCT04375319
Title: OCT Evaluation of Early Vascular Repair in Patients With Non ST Elevation Acute Coronary Syndrome (NSTE-ACS)
Acronym: EXPECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Third People's Hospital (Other)
Collaborators: Shandong Jiwei Medical Products Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-C-008-A07-V1.0
Record Dates: First submitted 2020-04-22; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Unstable Anginas; Non ST Segment Elevation Myocardial Infarction
Keywords: Optical Coherence Tomography; Drug Eluting Stents; EXCROSSAL
MeSH Terms: conditions — Angina, Unstable | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OCT guided 3-month follow-up group (Experimental): OCT guided the operation, and OCT reexamined 3 months after the operation to evaluate the vascular repair
  Interventions: Device: OCT
- 3-month follow-up group under the guidance of angiography (No Intervention): Coronary angiography guides the operation, OCT reexamination 3 months after operation to evaluate vascular repair
- 6-month follow-up group under the guidance of angiography (No Intervention): Coronary angiography guides the operation, OCT reexamination 6 months after operation to evaluate vascular repair

INTERVENTIONS:
Device: OCT — OCT can provide clear in vivo imaging and evaluate the vascular repair after stent implantation by measuring the optical echo of near-infrared light reflection
  Other Names: optical coherence tomography
  Arms: OCT guided 3-month follow-up group

SUMMARY:
This is a prospective study of a new generation of drug-eluting stent in the treatment of non ST elevation acute coronary syndrome (NSTE-ACS). The purpose of this study was to evaluate the extent of early vascular repair in NSTE-ACS patients after receiving the new generation of drug-eluting stents, and the value of OCT guided optimal implantation in further improving the target vascular endothelial repair, so as to provide the basis for early discontinuation of dual antiplatelet drugs (dapt) in NSTE-ACS patients and later large-scale randomized clinical research.This study is a prospective, multicenter, randomized controlled clinical study. Sixty patients with non ST elevation acute coronary syndrome (NSTE-ACS), including unstable angina and acute non ST elevation myocardial infarction, were enrolled in this study. After obtaining the written consent of the patients, the computer-generated random sequence table was randomly divided into three-month follow-up group (O3 group, n = 20), three-month follow-up group (A3 group, n = 20) and six-month follow-up group (A6 group, n = 20). Among them, the OCT guidance group needs to optimize the operation according to the examination results before and after the operation, while the contrast guidance group only conducts OCT examination collection after the operation. During the study period, all patients were given dual antiplatelet therapy (aspirin 100mg / D, clopidogrel 75mg QD or tegrilol 90mg bid). Sixty patients were followed up at 30 days, 3 months, 6 months and 1 year after stent implantation, and OCT was performed at 3 or 6 months after stent implantation, with the coverage rate of neointima as the main observation index. In this experiment, the independent OCT imaging laboratory, data management and Statistics Center, clinical endpoint determination Committee and clinical supervision organization collected, sorted, statistically analyzed and determined all relevant clinical and OCT imaging data. All the selected patients were followed up continuously within one year (telephone or outpatient follow-up) to observe the occurrence of adverse events.Primary end point: stent endometrial coverage measured by OCT (%)。

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled clinical trial, which will adopt the central randomized method based on computer system. When a patient signs the informed consent form and meets the inclusion criteria of the trial, and there is no exclusion criteria for randomization, the researcher fills in the randomization application form, and carries out randomization by landing on the randomization website randomization system. The computer system will automatically assign the randomization number and the corresponding treatment group according to the patient's situation. After obtaining the randomization results, the researcher should be in the randomization application form and the original The random number was recorded on the case and the patients were treated according to the group (Trial / control) assigned by the system.

The trial was carried out according to the following procedures: (1) signing informed consent; (2) case screening; (3) case selection; (4) The baseline OCT imaging was completed in the O3 group (including preoperative, intraoperative and postoperative use), and only OCT examination was performed in the A3 and A6 groups (not used to guide the optimization of PCI operation); (5) Follow up evaluation: ① OCT follow-up was conducted 3 or 6 months after the operation, and the imaging results were sent to the medical imaging analysis department for qualitative and quantitative evaluation and analysis; ② outpatient or telephone follow-up was conducted 1, 3, 6 and 12 months after the operation, and cardiovascular clinical events were recorded; The results of optical coherence tomography (OCT) in this study were evaluated by medical imaging analysis department. According to the standard procedure, the results of OCT imaging after stent implantation, 3 or 6 months after operation and any unexpected results are sent to the medical imaging analysis department, and the qualitative and quantitative evaluation analysis are completed by experienced image analysts. When the medical imaging analysis department evaluates the imaging results, it does not know whether the patients come from the experimental group or the control group, that is, they are always in a blind state. All calculation results were unblinded at the same time when the main end point data of the test were completed.

The task of data management and statistical analysis of this experiment will be undertaken by clinical research center of cardiovascular medicine of the third people's Hospital of Xuzhou City, and the statistical professionals will participate in the whole process of research design, implementation, data management and analysis and summary of test results. After the completion of the study plan and case report form, a statistical analysis plan will be made to complete the statistical analysis report.

The case report form (CRF) is filled in by the investigator, and each selected case must complete the CRF. After the completed case report form is reviewed by the supervisor, the first copy is transferred to the data administrator for data entry and management. After the first copy is handed over, the contents of the case report form will not be modified. The data administrator uses software to compile data entry program for data entry and management. In order to ensure the accuracy of the data, two data entry personnel shall independently enter and proofread the data in duplicate. For the questions in the case report form, the data administrator will send a query to the researcher by generating a question answer form (QF, query form), and contact the researcher through the supervisor to answer and return as soon as possible; the data administrator will modify, confirm and input the data according to the researcher's answers, and can send a QF again if necessary. After the data is reviewed and confirmed to be correct, the data management personnel, main researchers, statistical analysts, implementers and audit management personnel shall jointly review the data, and complete the final definition and judgment of the analysis population, and then the data administrator shall lock the database. Generally, the locked database or file cannot be changed. After the database is locked, submit it to the statistical analyst for statistical analysis.

During the clinical trial, the investigator of the hospital where the implementer is located and the investigator of the third people's Hospital of Xuzhou City will visit the research center regularly to ensure that all contents of the research scheme are strictly observed, and the original data are checked to ensure that the content of CRF is true, complete and correct.

Definition of adverse event: refers to any medical event, unexpected disease or injury, or unfortunate clinical sign that occurs to the subject, user or other personnel during the period from the time when the patient agrees to participate in the study to the time when the patient no longer participates in the study, whether related to the medical device under study or not.

Severity of adverse events: ① mild: no impact on daily activities; ② moderate: impact on daily activities; ③ severe: loss of ability of daily activities.

Response measures for adverse events: all adverse events occurred during the study must be recorded in the adverse event table truthfully. The researchers should give targeted treatment and follow-up until the symptoms disappear or stable.

Serious adverse events: serious adverse events refer to the events that need hospitalization treatment, prolong hospitalization time, disability, affect work ability, endanger life or death, cause congenital malformation, etc. during the clinical trial. In case of serious adverse events during the study, whether related to the trial dose or not, appropriate treatment measures must be taken immediately, and at the same time, they shall be reported to the administrative departments, implementers and clinical supervisors of the main researchers, the ethics committee of the clinical research responsible unit, the provincial and Municipal Health and family planning committees, etc. by telephone or fax within 24 hours after being informed, and The serious adverse event record form shall be submitted within 24 hours after learning.

Statistical analysis method:

Descriptive analysis: composition ratio is used to describe counting data, mean, standard deviation, maximum value and minimum value are used to describe measuring data, mean, standard deviation, maximum value, minimum value, median, 25th and 75th quantiles are used to describe non normal distribution data.

Baseline demographic analysis: when the theoretical frequency in the four grid table is less than 5, Fisher's exact probability method is used; group t test (two groups) or variance analysis (multiple groups) are used for the comparison of normal distribution measurement data; Wilcoxon rank sum test is used for the comparison between groups.

Efficacy analysis: paired t-test was used for comparison in normal distribution measurement group, and Wilcoxon rank sum test was used for comparison in non normal distribution measurement group. After the homogeneity of variance between the two groups was tested, the covariance analysis of adjusted center effect and baseline effect was used, and the least mean square of dependent variable, the least mean square of group, and 95% confidence interval were given to test the zero hypothesis; the CMH (Cochran mantel Haenszel) χ 2 test of adjusted center effect was used for the inter group comparison of count data.

Safety evaluation: according to the experimental group and the control group, describe the number and proportion of normal cases before and after treatment. Adverse events were described by the number and incidence of adverse events, and the proportion was tested by χ 2 test or Fisher exact probability method. At the same time, detailed description of all adverse events in each group, the specific performance, degree and the relationship with the dosage.

All statistical analysis will be performed at the bilateral 0.05 significance level. Sas9.13 statistical software is used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant female aged 18-80;
* Patients with unstable angina or acute non ST segment elevation myocardial infarction have been diagnosed clinically;
* The target lesions are primary and in situ coronary lesions. If there are multiple target lesions, they must be located in different epicardial vessels;
* The total length of each target lesion is ≤ 40mm, and the diameter of the target vessel is 2.5mm-4.5mm (visual method);
* The stenosis degree of target lesion ≥ 70% or the stenosis degree of target lesion with evidence of myocardial ischemia ≥ 50% (visual method);
* Each patient is allowed to implant at most 3 homostents (except for salvage implantation of additional stents), and each target lesion is allowed to implant at most 2 homostents;
* Patients with indication of coronary artery bypass surgery;
* Patients who can understand the purpose of this trial, voluntarily participate in and sign the informed consent, have good compliance after discharge, take medicine on time, and are willing to receive optical coherence tomography (OCT) examination and clinical follow-up.

Exclusion Criteria:

* Any acute ST segment elevation myocardial infarction within 1 month;
* Chronic total occlusion (preoperative Timi Grade 0 blood flow), severe left main coronary artery disease, long disease (disease length > 40mm), bifurcated disease with double stenting, diameter of disease vessel > 4.5mm, incomplete optical coherence tomography (OCT) at the lesion site or the disease is not suitable for OCT imaging, bypass vessel disease, visible thrombus in the target vessel, concurrent infection or other inflammatory diseases;
* Severe calcification and tortuosity can not be successfully pre dilated, which is not suitable for stent delivery and expansion;
* Restenosis in stent;
* Patients who had implanted any brand of stent in one year, those who had the possibility of reoperation in one year, and those who had implanted stent for more than one year;
* Hemodynamics or respiratory and circulatory instability have been demonstrated, such as cardiogenic shock, severe heart failure (NYHA III and above) or left ventricular ejection fraction < 40% (ultrasound or left ventriculography);
* The renal function was damaged before operation: EGFR < 60ml / (min · 1.73m2) or serum creatinine > 2.5mg/dl (178 μ mol / L);
* Patients with bleeding tendency, history of active peptic ulcer, history of cerebral hemorrhage or subretinal hemorrhage, history of stroke within half a year, contraindications of antiplatelet agents and anticoagulants cannot receive anticoagulant treatment;
* Allergic to aspirin, clopidogrel or tegrelol, statins, heparin, contrast agents, polymers, zoltamox and metals;
* The life expectancy of patients is less than 12 months;
* Those who have participated in clinical trials of other drugs or medical devices before being selected but failed to reach the time limit of main research end point;
* The researcher judges that the patient's compliance is poor and is unable to complete the study as required, unwilling or unable to provide written informed consent;
* Heart transplant patients;
* There are unstable arrhythmias, such as high-risk ventricular premature beats and ventricular tachycardia;
* Because the tumor needs chemotherapy within 30 days;
* Have immunosuppressive, autoimmune diseases, plan or are receiving immunosuppressive treatment;
* Patients who need to stop aspirin, clopidogrel or tegrilol due to selective surgery within half a year;
* Blood routine examination showed that platelet count was lower than 100 × 10∧9/ L, or higher than 700 × 10∧9 / L, leukocyte was lower than 3 × 10∧9 / L, and liver diseases (such as hepatitis) were diagnosed or suspected;
* The patient had diffuse peripheral vascular disease and could not use 6F catheter.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Stent endometrial coverage measured by OCT | 3 to 6 months after operation
  Patients were randomly assigned to the 3-month or 6-month follow-up group。According to the randomized group, Oct reexamination was carried out at 3 or 6 months after the operation to evaluate the stent endometrial coverage rate。

SECONDARY OUTCOMES:
Poor adherence rate of stent wire during follow-up | 3 to 6 months after operation
  Patients were randomly assigned to the 3-month or 6-month follow-up group。At 3 or 6 months after the operation, Oct reexamination was carried out to observe and record the bad rate of stent wire sticking to the wall
minimum and average lumen area, the minimum stent area and the average stent area | 3 to 6 months after operation
  Patients were randomly assigned to the 3-month or 6-month follow-up group。OCT measures theminimum and average lumen area, the minimum stent area and the average stent area,The unit is:mm^2
Minimum stent diameter and average stentdiameter,minimum lumen diameter and average lumen diameter | 3 to 6 months after operation
  Patients were randomly assigned to the 3-month or 6-month follow-up group。OCT measures the Minimum stent diameter and average stentdiameter,minimum lumen diameter and average lumen diameter,The unit is:mm
Covering thickness of scaffold surface structure | 3 to 6 months after operation
  Patients were randomly assigned to the 3-month or 6-month follow-up group。The high resolution of OCT may provide a detailed analysis and evaluation of whether the stent surface has endometrial coverage and the extent of tissue coverage, and record and analyze the minimum and average values.
Vascular repair index | 3 to 6 months after operation
  Patients were randomly assigned to the 3-month or 6-month follow-up group。At 3 or 6 months after operation, the patients were reexamined by OCT, and the vascular repair index was observed and recorded，The higher the vascular repair index, the better the result
cardiovascular death | 30 days, 3 months, 6 months and 1 year after operation
  Observe and record the number of cardiac deaths at 30 days, 3 months, 6 months and 1 year
Nonfatal myocardial infarction | 30 days, 3 months, 6 months and 1 year after operation
  Observe and record the number of Nonfatal myocardial infarction at 30 days, 3 months, 6 months and 1 year
All revascularization | 30 days, 3 months, 6 months and 1 year after operation
  Observe and record the number of All revascularization at 30 days, 3 months, 6 months and 1 year
Target lesion revascularization | 30 days, 3 months, 6 months and 1 year after operation
  Observe and record the number of Target lesion revascularization at 30 days, 3 months, 6 months and 1 year
Target vessel revascularization | 30 days, 3 months, 6 months and 1 year after operation
  Observe and record the number of Target vessel revascularization at 30 days, 3 months, 6 months and 1 year
Stent thrombosis | 30 days, 3 months, 6 months and 1 year after operation
  Observe and record the number of Stent thrombosis at 30 days, 3 months, 6 months and 1 year

OTHER OUTCOMES:
Blood lipid level：Include LDL、HDL、LDL 、HDL | Before surgery 、One day after operation、 3 months after operation、 6 months after operation
  Observe and record these indicators according to time nodes，The unit is:mmol/L
Biological indicators：hs-CRP（mg/L） | Before surgery 、One day after operation、 3 months after operation、 6 months after operation
  Observe and record these indicators according to time nodes,Comparative 。analysis of changes in time nodes。The unit is:mg/L
Biological indicators：PTX-3、VCAM-1、MMP-9 | Before surgery 、One day after operation、 3 months after operation、 6 months after operation
  Observe and record these indicators according to time nodes,Comparative analysis of changes in time nodes

CONTACTS AND LOCATIONS:
Overall Officials: yaojun zhang, Doctorate, Principal Investigator — Head of Cardiology Department of Xuzhou Third People's Hospital
Locations (2):
- China (2):
  - Xuzhou Third People's Hospital, Xuzhou, Jiangsu
  - Peixian Guotai hospital, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No
It's not decided whether to share

REFERENCES:
- [Result] Iliescu CA, Cilingiroglu M, Giza DE, Rosales O, Lebeau J, Guerrero-Mantilla I, Lopez-Mattei J, Song J, Silva G, Loyalka P, Paixao ARM, Yusuf SW, Perin E, Anderson VH, Marmagkiolis K. "Bringing on the light" in a complex clinical scenario: Optical coherence tomography-guided discontinuation of antiplatelet therapy in cancer patients with coronary artery disease (PROTECT-OCT registry). Am Heart J. 2017 Dec;194:83-91. doi: 10.1016/j.ahj.2017.08.015. Epub 2017 Aug 23. PMID 29223438
- [Result] Shlofmitz E, Garcia-Garcia HM. The Role of OCT Guidance for Antiplatelet Therapy. Cardiovasc Revasc Med. 2018 Oct;19(7 Pt A):733-734. doi: 10.1016/j.carrev.2018.09.015. No abstract available. PMID 30420093
- [Result] Laine M, Dabry T, Combaret N, Motreff P, Puymirat E, Paganelli F, Thuny F, Cautela J, Peyrol M, Mancini J, Lemesle G, Bonello L. OCT Analysis of Very Early Strut Coverage of the Synergy Stent in Non-ST Segment Elevation Acute Coronary Syndrome Patients. J Invasive Cardiol. 2019 Jan;31(1):10-14. doi: 10.25270/jic/18.00274. Epub 2018 Nov 11. PMID 30418164
- [Result] Won H, Shin DH, Kim BK, Mintz GS, Kim JS, Ko YG, Choi D, Jang Y, Hong MK. Optical coherence tomography derived cut-off value of uncovered stent struts to predict adverse clinical outcomes after drug-eluting stent implantation. Int J Cardiovasc Imaging. 2013 Aug;29(6):1255-63. doi: 10.1007/s10554-013-0223-9. Epub 2013 Apr 25. PMID 23615849
- [Result] Adriaenssens T, Joner M, Godschalk TC, Malik N, Alfonso F, Xhepa E, De Cock D, Komukai K, Tada T, Cuesta J, Sirbu V, Feldman LJ, Neumann FJ, Goodall AH, Heestermans T, Buysschaert I, Hlinomaz O, Belmans A, Desmet W, Ten Berg JM, Gershlick AH, Massberg S, Kastrati A, Guagliumi G, Byrne RA; Prevention of Late Stent Thrombosis by an Interdisciplinary Global European Effort (PRESTIGE) Investigators. Optical Coherence Tomography Findings in Patients With Coronary Stent Thrombosis: A Report of the PRESTIGE Consortium (Prevention of Late Stent Thrombosis by an Interdisciplinary Global European Effort). Circulation. 2017 Sep 12;136(11):1007-1021. doi: 10.1161/CIRCULATIONAHA.117.026788. Epub 2017 Jul 18. PMID 28720725
- [Result] Zaman A, de Winter RJ, Kogame N, Chang CC, Modolo R, Spitzer E, Tonino P, Hofma S, Zurakowski A, Smits PC, Prokopczuk J, Moreno R, Choudhury A, Petrov I, Cequier A, Kukreja N, Hoye A, Iniguez A, Ungi I, Serra A, Gil RJ, Walsh S, Tonev G, Mathur A, Merkely B, Colombo A, Ijsselmuiden S, Soliman O, Kaul U, Onuma Y, Serruys PW; TALENT trial investigators. Safety and efficacy of a sirolimus-eluting coronary stent with ultra-thin strut for treatment of atherosclerotic lesions (TALENT): a prospective multicentre randomised controlled trial. Lancet. 2019 Mar 9;393(10175):987-997. doi: 10.1016/S0140-6736(18)32467-X. Epub 2019 Feb 28. PMID 30827782
- [Result] Lee BK, Kim JS, Lee OH, Min PK, Yoon YW, Hong BK, Shin DH, Kang TS, Kim BO, Cho DK, Jeon DW, Woo SI, Choi S, Kim YH, Kang WC, Kim S, Kim BK, Hong MK, Jang Y, Kwon HM. Safety of six-month dual antiplatelet therapy after second-generation drug-eluting stent implantation: OPTIMA-C Randomised Clinical Trial and OCT Substudy. EuroIntervention. 2018 Mar 20;13(16):1923-1930. doi: 10.4244/EIJ-D-17-00792. PMID 29104179
- [Derived] Zhu YX, Liang L, Parasa R, Li Z, Li Q, Chang S, Ma WR, Feng SL, Wang Y, Xu B, Bourantas CV, Zhang YJ. Early vascular healing after neXt-generation drug-eluting stent implantation in Patients with non-ST Elevation acute Coronary syndrome based on optical coherence Tomography guidance and evaluation (EXPECT): study protocol for a randomized controlled trial. Front Cardiovasc Med. 2023 Feb 23;10:1003546. doi: 10.3389/fcvm.2023.1003546. eCollection 2023. PMID 36910518